CLINICAL TRIAL: NCT06312098
Title: The Study on Perioperative Factors Affecting Postoperative Outcomes in Patients Who Underwent Adult Liver Transplantation
Brief Title: Perioperative Factors and Living Donor Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Min Suk Chae (Other)
Responsible Party: Sponsor-Investigator, Min Suk Chae, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: KC21RISI0576
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Liver Transplant Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no-remote ischemic preconditioning group: patients who did not receive remote ischemic preconditioning
- paired remote ischemic preconditioning group: patients who receive remote ischemic preconditioning
  Interventions: Other: remote ischemic preconditioning (RIPC)

INTERVENTIONS:
Other: remote ischemic preconditioning (RIPC) — After induction of anesthesia, the paired RIPC group took the RIPC intervention on the upper arm in the lateral position. The RIPC intervention was applied using a manual cuff inflator, which consisted of three cycles of 5-min inflation of the blood pressure cuff (to 250 mmHg, or to 50 mmHg higher than the preoperative SBP), followed by 5-min deflation of the cuff. In the no-RIPC group, a blood pressure cuff was also applied on the upper arm but was not inflated.
  Groups: paired remote ischemic preconditioning group

SUMMARY:
Liver transplant surgery is one of the treatments provided to patients suffering from end-stage liver disease, and has a successful treatment prognosis. However, it is clear that patient management before, during, and after surgery is a difficult task for medical staff due to the complex clinical and pathological problems of end-stage liver disease. Moreover, the complex surgical technique of the liver transplant surgery itself and the severe hemodynamic fluctuations and multi-organ dysfunction that patients experience during the surgery have been shown to have a tremendous impact on the patient's prognosis after surgery.

A study on which clinical, laboratory, and hemodynamic factors experienced by patients during the perioperative period, including before, during, and after surgery, affect the survival rate of patients and transplanted organs. will definitely be helpful in the treatment of patients suffering from end-stage liver disease.

ELIGIBILITY:
Inclusion Criteria:

* adults
* elective surgery
* American Society of Anesthesiologists (ASA) physical status classification system I, II, III

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification system IV, V

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from adult patients undergoing elective living donor liver transplantation at Seoul St. Mary's Hospital were retrospectively collected with the electronic medical record system.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postreperfusion syndrome | during surgery
  mean blood pressure decreases by 30% based on the value on preoperative day

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during this study are available from the corresponding author on reasonable request.